CLINICAL TRIAL: NCT01888406
Title: Targeting Binge Eating to Prevent Weight Gain in College Students
Brief Title: Binge Eating Self-help Treatment for University Students
Acronym: BEST4US
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Francine Rosselli (Other)
Collaborators: Wesleyan University (Other)
Responsible Party: Sponsor-Investigator, Francine Rosselli, Visting Scholar, Dept of Psychology; Co-Investigator, BEST4US, Wesleyan University
Organization: Wesleyan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R15DK092768-O1A1; 1R15DK092768 (NIH)
Record Dates: First submitted 2013-06-20; First posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Obesity; Binge Eating Disorder
Keywords: Obesity; Weight gain prevention; Eating disorder; Binge eating
MeSH Terms: conditions — Obesity; Binge-Eating Disorder; Feeding and Eating Disorders; Bulimia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guided Self-Help (Experimental): Participants receive self-help materials, including a book (Overcoming Binge Eating by C. Fairburn, handouts, and online resources. In addition, participants receive 8 individual sessions with a peer coach who supports participants in working the self-help program.
  Interventions: Behavioral: Guided Self-Help
- Pure Self-Help (Other): Participants receive self-help materials, including a book (Overcoming Binge Eating by C. Fairburn, handouts, and online resources.
  Interventions: Behavioral: Pure Self-Help

INTERVENTIONS:
Behavioral: Guided Self-Help
  Arms: Guided Self-Help
Behavioral: Pure Self-Help
  Arms: Pure Self-Help

SUMMARY:
BEST4US compares the effectiveness of two forms of self-help interventions that target college students, ages 18 years to 22 years, who report binge eating. The overall question is whether one or the other format will prevent excess weight gain and lead to differences in eating behaviors. The two formats are (1) "pure self-help" (receipt of a self-help program via book form or online texts) and (2) a combination of the self-help program and guidance provided by a trained peer coach over the course of 8 weekly sessions.

ELIGIBILITY:
Inclusion Criteria:

* binge eating episodes at least once per week in the past 28 days
* 18 to 22 years old
* full-time student at Wesleyan University (Middletown, CT, USA) or Manchester Community College (Manchester, CT, USA)

Exclusion Criteria:

* purging more than once per week in the past three months
* BMI less than 18 or greater than/equal to 40
* currently pregnant
* severe depressive symptoms or suicidality

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
BMI | Baseline, post-intervention (8-week), and 6-month follow-up
  The primary outcome measure is change in BMI from randomization. Height and weight will be measured by study staff at the baseline visit using a stadiometer (collecting height measures twice and reporting the average) and a calibrated scale (light clothing, street shoes removed). BMI will be calculated as weight in kilograms divided by height in squared centimeters. Weight will be re-measured at 8 week- and 6 month assessments. BMI change is a primary-, and incidence of obesity (i.e., obesity onset since baseline, BMI > 30) is a secondary outcome variable. While we assess weight at the post-treatment assessment, the key question of our study is whether the intervention will reduce excess weight gain at 6-month follow-up.

SECONDARY OUTCOMES:
Cessation of Binge Eating | Baseline, post-intervention (8-week), and 6-month follow-up
  Binge eating is assessed by clinical interview using an abbreviated version of the Eating Disorders Examination (EDE-16e) at baseline, post-treatment (8-week), and 6-month follow-up. Specifically, the EDE sections on 7-day meal patterns, overeating episodes, and the frequency of inappropriate compensatory behaviors will be administered. The key question of our study is whether the intervention will eliminate binge eating at 6-month follow-up (no reported binge eating episodes in the 28 days prior to the 6-month follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Striegel, PhD, Principal Investigator — Wesleyan University; Francine Rosselli, PhD, Study Director — Manchester Community College
Locations (2):
- United States (2):
  - Manchester Community College Department of Psychology, Manchester, Connecticut
  - Wesleyan University Department of Psychology, Middletown, Connecticut